CLINICAL TRIAL: NCT03585062
Title: Clinical Trial of Neoadjuvant Chemotherapy With S1 Plus Paclitaxel-albumin in Patients With Unresectable Locally Advanced Pancreatic Cancer
Brief Title: Trial of Neoadjuvant Chemotherapy With S1 Plus Paclitaxel-albumin on Pancreatic Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The paclitaxel-albumin halt production.
Sponsor: Zhejiang Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Yi-Ping Mou, Vice Present of Zhejiang Provincial People's Hospital, Zhejiang Provincial People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017KY007
Record Dates: First submitted 2018-01-08; First posted 2018-07-12 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Pancreatic Cancer; Neoadjuvant Chemotherapy
Keywords: S-1; Paclitaxel-albumin; Unresectable Pancreatic Cancer; Neoadjuvant chemotherapy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — S 1 (combination); gimeracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- S-1 combined with Paclitaxel-albumin (Experimental): S-1 combined with Paclitaxel-albumin S-1:40~60mg bid, day 1~14 (S-1: BSA <1.25m2, 40mg bid , 1.25m2 ≤ BSA ≤1.5m2, 50mg bid, BSA>1.5m2, 60mg bid， for 2 weeks, rest a week) Paclitaxel-albumin: 125 mg/m2, intravenous infusion for 30 minutes, Day1 and Day 8.
  Interventions: Drug: S1,; Drug: Paclitaxel-albumin

INTERVENTIONS:
Drug: S1, — S-1 is a combination of tegafur, gimeracil and oteracil at a molar ratio of 1:0.4:1, and is a new oral fluoropyrimidine anticancer agent shown to be effective for pancreatic cancer. cancer
  Other Names: Gimeracil and Oteracil Porassium Capsules
Drug: Paclitaxel-albumin — Paclitaxel-albumin is a drug which showed a survival benefit in Pancreatic Cancer when combined with S1

SUMMARY:
The study is to evaluate the R0 resection rate of patients with unresectable locally advanced pancreatic cancer ,after treated with S-1 plus Paclitaxel-albumin as neoadjuvant chemotherapy protocols

DETAILED DESCRIPTION:
BACKGROUND:

1. The incidence of pancreatic cancer in China has been increasing rapidly in recent years，but most of the pancreatic cancer patients are unresectable, whose median survival time were only 6~9 months.
2. Studies have shown that neoadjuvant therapy improves the quality of surgery in patients with pancreatic cancer，and prolong their life.
3. S-1 is a new generation of oral fluorouracil derivatives ,S-1 single drug as an adjuvant therapy for resectable pancreatic cancer is better than gemcitabine, and has less side effects than gemcitabine. Protein bound paclitaxel is a novel paclitaxel combined of paclitaxel and albumin by nanotechnology , which can extend free survival in patients with advanced pancreatic cancer with less side effects than gemcitabine. So S-1 combined with Paclitaxel-albumin is expected to play an important role in neoadjuvant chemotherapy in Pancreatic cancer, and may improve the rate of R0 resection in patients with unresectable locally advanced pancreatic.

STUDY DESIGN:

S-1 combined with Paclitaxel-albumin

1. S-1:40~60mg bid, day 1~14 (S-1: BSA (Body surface area)<1.25m2, 40mg bid , 1.25m2 ≤ BSA ≤1.5m2, 50mg bid, BSA>1.5m2, 60mg bid),2 weeks and rest for 1 weeks.
2. Paclitaxel-albumin: 125 mg/m2, intravenous infusion for 30 minutes, Day1 and Day 8.

Repeat every three weeks. for 6 cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed invasive ductal adenocarcinoma of pancreas by histology
2. Evaluated as CT4N0M0 pancreatic cancer patients by Image testing
3. Adults age from 18-80 years old
4. No history of pancreatic resection or pancreatic cancer
5. ECOG score 0-1; can be orally administered
6. No distant metastasis or malignant ascites
7. Relatively good liver、 kidney、heart、hematology function. Baseline blood routine and biochemical indexes of the subjects meet the following criteria: hemoglobin ≥90g/L;absolute neutrophil count(ANC)≥3.5×109/L；Platelet≥100×109/L;prothrombin time ≤1.8;partial thromboplastin time ≤1.8; ALT≤102U/L、AST≤95U/L; ALP≤2.5 times the upper limits of normal; Serum total bilirubin≤2.5 g/dL(total bilirubin ≤1.5 times the upper limit of normal (ULN)；Serum creatinine≤2.0 mg/dL； creatinine clearance rate >50 ml/min
8. Sign the Informed consent -

Exclusion Criteria:

1. Woman in pregnant or lactation period
2. Woman of childbearing age who was positive at baseline pregnancy test or did not have pregnancy tests.Menopausal women must have menopause for at least 12 months before they think they are free of pregnancy.
3. Men and women who had sexual life (Fertility possibility) were reluctant to have contraception during the study period.
4. Patients with the history of other malignant diseases in the past 5 years, except for cured skin cancer and cervical carcinoma in situ.
5. Patients of uncontrolled epilepsy, central nervous system diseases or history of mental disorders, should be judged by the researchers whether their clinical severity hinder the signature of the informed consent or influenced patients'compliance with oral medications
6. Clinically serious (i.e. activity) heart disease, such as symptomatic coronary heart disease , New York Heart Association (NYHA) class II or more serious congestive heart failure or serious arrhythmia which need drug intervention, or have a history of MI within the last 12 months.
7. Patients with upper gastrointestinal obstruction or Abnormal physiological function or Malabsorption syndrome, which may affect the absorption of S-1.
8. Organ transplant patients who need immunosuppressive therapy
9. Patients with Serious uncontrolled repeated infection or other serious uncontrolled Concomitant disease.
10. Patient that is lack of dihydropyrimidine dehydrogenase (DPD)
11. Allergic to any of the drug ingredients in this study
12. participate in other clinical trials within 4 weeks before randomization -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
R0 resection rate | one week After the operation
  Evaluate the R0 resection rate of S-1 combined with Paclitaxel-albumin as neoadjuvant chemotherapy in patients with unresectable locally advanced pancreatic cancer

SECONDARY OUTCOMES:
The objective remission rate (ORR) | at the end of cycle 6 of the neoadjuvant chemotherapy((each cycle is 21 days)
  Evaluate the objective remission rate (ORR) of S-1 combined with Paclitaxel-albumin as neoadjuvant chemotherapy in patients with unresectable locally advanced pancreatic cancer
The disease free survival (DFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first,assessed up to 60 months. Progressing should be confirmed by imaging examination or histology / cytology examination.
  Evaluate the disease free survival (DFS) of S-1 combined with Paclitaxel-albumin as neoadjuvant chemotherapy in patients with unresectable locally advanced pancreatic cancer
The 2 year and 5 year survival rate | 2 years and 5 years after treatment
  Evaluate the 2 year and 5 year survival rate of S-1 combined with Paclitaxel-albumin as neoadjuvant chemotherapy in patients with unresectable locally advanced pancreatic cancer
The quality of life | Questionnaire at baseline, and then 1-2 days before each cycle of treatment(each cycle is 21 days, for a total of 6 cycles.). During follow-up period after treatment, questionnaire every 6 months, up to 2 years.
  Assess the quality of life in pancreatic cancer according to EORTC QLQ-PAN26(European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Pancreas 26).For each assessment item, there are four options, scores are as 1,2,3,4. Each score corresponds to a physical condition. Then have the total score for each patient. The total score range from 26-104, the higher the score, the poorer the quality of life is.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang procincial people's hospital, Hanzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel R, Naishadham D, Jemal A. Cancer statistics, 2013. CA Cancer J Clin. 2013 Jan;63(1):11-30. doi: 10.3322/caac.21166. Epub 2013 Jan 17. PMID 23335087
- [Background] Jemal A, Bray F, Center MM, Ferlay J, Ward E, Forman D. Global cancer statistics. CA Cancer J Clin. 2011 Mar-Apr;61(2):69-90. doi: 10.3322/caac.20107. Epub 2011 Feb 4. PMID 21296855
- [Background] Witkowski ER, Smith JK, Tseng JF. Outcomes following resection of pancreatic cancer. J Surg Oncol. 2013 Jan;107(1):97-103. doi: 10.1002/jso.23267. Epub 2012 Sep 18. PMID 22991309
- [Background] Neoptolemos JP, Stocken DD, Friess H, Bassi C, Dunn JA, Hickey H, Beger H, Fernandez-Cruz L, Dervenis C, Lacaine F, Falconi M, Pederzoli P, Pap A, Spooner D, Kerr DJ, Buchler MW; European Study Group for Pancreatic Cancer. A randomized trial of chemoradiotherapy and chemotherapy after resection of pancreatic cancer. N Engl J Med. 2004 Mar 18;350(12):1200-10. doi: 10.1056/NEJMoa032295. PMID 15028824